CLINICAL TRIAL: NCT07216430
Title: A Phase 2 Study Evaluating the Safety and Efficacy of Whole-Cell Pneumococcal Vaccine (wSp) in Reducing Nasopharyngeal Colonization by Streptococcus Pneumoniae in Young Children.
Brief Title: Safety and Efficacy of wSp Vaccine in Young Children
Acronym: wSp005
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Serum Life Science Europe GmbH (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Rochester General Hospital (Other); Serum Institute of India Pvt. Ltd. (Industry); Alira Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: wSp-US-2.03AOM; 1U01AI172733-01A1 (NIH)
Record Dates: First submitted 2025-09-25; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Otitis Media (AOM)
MeSH Terms: conditions — Otitis Media | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the person administering the investigational product will be unmasked. This person does not perform any other participant-related tasks in the clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2x 1 mg wSp vaccine (Experimental): Intramuscular (IM) injections of 0.5 mL containing 1 mg of total protein
  Interventions: Biological: wSp vaccine
- 2x 0.5 mL saline (Placebo Comparator): Intramuscular (IM) injections of 0.5 mL saline
  Interventions: Biological: Saline (0.9% NaCl)

INTERVENTIONS:
Biological: wSp vaccine — wSp vaccine will be administered as intramuscular (IM) injections of 0.5 mL (thus 1 mg total protein). wSp vaccine is supplied as single-dose glass vials in saline (0.9% sodium chloride) at 2 mg protein/mL, with aluminum hydroxide at 1.2 mg elemental Al/mL. Dose 1 will be given in the left thigh at 7 months of age, and dose 2 will be given in the right thigh at 9 months of age.
  Other Names: SPWCV; PATH-wSP
  Arms: 2x 1 mg wSp vaccine
Biological: Saline (0.9% NaCl) — Saline will be administered as intramuscular (IM) injections of 0.5 mL. Dose 1 will be given in the left thigh at 7 months of age and dose 2 will be given in the right thigh at 9 months of age.
  Arms: 2x 0.5 mL saline

SUMMARY:
The goal of this clinical trial is to evaluate whether the wSp vaccine can prevent nasopharyngeal colonization by pneumococcal bacteria in healthy young children who have received routine PCV20 vaccination.

The main questions it aims to answer are:

Does wSp vaccine reduce pneumococcal colonization in the nose? Does wSp vaccine safely stimulate the immune system to produce antibodies and protective immune responses?

Researchers will compare children receiving two injections of wSp vaccine to those receiving saline placebo to see if wSp vaccine reduces colonization and boosts immunity.

Participants will:

Receive two injections of either wSp or saline at 7 and 9 months of age. Have blood samples taken at 6 and 12 months to measure immune responses. Have nasal swabs collected at several time points and during infections from 6-24 months.

Be monitored for ear infections, respiratory illnesses, and other pneumococcal-related infections.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female who is 6 months (+/- 30 days) of age at time of enrollment
2. Healthy subject as established by medical history and clinical examination before entering into the study.
3. Received 3 doses of PCV-20.
4. Written informed consent obtained from the subject's parent/legal guardian.
5. Parent/legal guardian able and willing to bring subject to all study visits.

Exclusion Criteria:

1. Has a history of invasive pneumococcal disease (positive blood culture and/or positive cerebrospinal fluid culture).
2. Known or suspected impairment of immunological function, based on medical history and physical examination.
3. Has a history of congenital or acquired immunodeficiency.
4. Chronic administration (defined > 14 consecutive days) of immunosuppressants or other immune-modifying drugs, or during the study period.
5. Prior receipt since birth of immunoglobulins and/or any blood products or planned administration during the study period.
6. Expected to receive systemic corticosteroids within 14 days prior to any dose of study vaccine.
7. External auditory canal atresia/stenosis.
8. Has known or history of functional or anatomic asplenia.
9. Has a bleeding disorder in which intramuscular vaccination would be contraindicated.
10. Participation in another investigational or interventional trial within the 28-day period before enrollment and during the conduct of the study. Participation in observational studies is permitted.
11. Direct descendant (child or grandchild) of study site personnel.

    Temporary exclusion criteria

    For day of vaccination:
12. Fever (transcutaneous temperature ≥38.0°C) or acute illness
13. Has received systemic corticosteroids (equivalent of prednisone > 0.5 mg/kg/day or equivalent) and not completed this course of treatment at least 30 days prior to the study vaccination. Inhaled, topical, and ophthalmic steroids are allowed.

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Occurrences of Streptococcus pneumoniae in the nasopharynx | 3, 6, 9 and 15 months after second dosing, if healthy, and 14 days through 15 months after second dosing at the time of AOM, LRTI, and/or URTI episodes
  Occurrence of a culture-confirmed S. pneumoniae of differing serotypes in the nasopharynx (as defined by isolation of S. pneumoniae from NP samples)
  * at four healthy visits, child age 12, 15, 18 and 24 months old and/or
  * 14 days after second vaccine dose through 24 months of age, at AOM, LRTI, and URTI visits throughout study participation.

SECONDARY OUTCOMES:
Occurrence of new serotype of Streptococcus pneumoniae in the nasopharynx during viral upper respiratory infection at onset of acute otitis media | between 14 days after the second dose of vaccine and 24 months of age
  Occurrence of a culture-confirmed new serotype of S. pneumoniae in the nasopharynx during viral URI at onset of AOM (as defined by isolation of S. pneumonia of differing serotypes from NP samples) between 14 days after the second dose of vaccine and 24 months of age

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Western New York Geneva Pediatrics, Rochester, New York
  - Bay Creek Pediatrics, Rochester, New York
  - Rochester Medical Group General Pediatric Associates, Rochester, New York
  - Panorama Pediatrics, Rochester, New York

IPD SHARING:
Plan to Share IPD: No